CLINICAL TRIAL: NCT06095128
Title: An Open-Label, Phase 4, Single-Arm, Multicenter Study to Evaluate the Induction of Response and Remission of Vedolizumab Dual Targeted Therapy With Tofacitinib in Adult Patients With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of Vedolizumab With Tofacitinib in Adults With Ulcerative Colitis (UC)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vedolizumab-4054
Record Dates: First submitted 2023-10-18; First posted 2023-10-23 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis
Keywords: Drug Therapy
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab; tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vedolizumab 300 mg + Tofacitinib 10 mg (Experimental): Participants will receive Vedolizumab 300 mg, intravenous (IV) infusion, at Week 0, Week 2 and Week 6 along with Tofacitinib 10 mg, tablets, orally, twice daily from Week 0 to Week 8. Participants with clinical response at Week 8 will transition to receive vedolizumab 300 mg IV infusion every 8 weeks (Q8W) through Week 46.
  Interventions: Drug: Vedolizumab; Drug: Tofacitinib

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab IV infusions
  Other Names: Entyvio; MLN0002
Drug: Tofacitinib — Tofacitinib Tablets
  Other Names: Xeljanz; CP-690; CP-550

SUMMARY:
The main aim of this study is to learn about the effect of treatment with vedolizumab IV (vedolizumab) together with tofacitinib in adults with moderate and severe ulcerative colitis (UC). Another aim is to learn about treatment with Vedolizumab alone after the double treatment.

All participants will receive vedolizumab together with tofacitinib for 8 weeks and will be checked for response. Participants who show a response to the treatment after 8 weeks will be treated with vedolizumab alone for an additional 44 weeks.

Each participant will be followed up for at least 26 weeks after the last dose of vedolizumab.

DETAILED DESCRIPTION:
The drugs being tested in this study are called Vedolizumab and Tofacitinib. Vedolizumab and Tofacitinib dual targeted therapy is being tested to treat people with moderate to severe ulcerative colitis (UC) who have experienced inadequate response, loss of response or intolerance to no more than 2 prior tumor necrosis factor (TNF) antagonists. This study will look at the clinical remission in people who take Vedolizumab and Tofacitinib dual targeted therapy.

The study will enroll approximately 65 patients. All the participants will be enrolled in a single treatment group to receive dual targeted treatment with Vedolizumab and Tofacitinib for the first 8 weeks:

Vedolizumab 300 mg + Tofacitinib 10 mg

Only those participants who show a clinical response at Week 8 will transition to Vedolizumab monotherapy for 44 weeks.

This multi-center trial will be conducted in the United States and Canada. The overall duration of the study is up to 76 weeks. Participants will be followed up for 26 weeks after the last dose of the study drug for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Has a confirmed diagnosis of UC established at least 3 months prior to screening, by clinical and endoscopic evidence and corroborated by a histopathology report.
2. Has moderately to severely active UC as determined by a complete Mayo score [including physician's global assessment (PGA)] of 6 to 12 with a rectal bleeding subscore ≥1 and a centrally assessed endoscopic subscore ≥2 at screening.
3. Has evidence of UC extending proximally to the rectum [≥15 centimeter (cm) of involved colon].
4. Participants with extensive colitis or pancolitis of >8 years duration or left sided colitis >12 years duration must have documented evidence that a surveillance colonoscopy was performed within 12 months of the initial screening visit.
5. Participants with a family history of colorectal cancer, personal history of increased colorectal cancer risk, age >50 years, or other known risk factors must be up to date on colorectal cancer surveillance.
6. Has demonstrated an inadequate response to, loss of response to, or intolerance to at least 1, but no more than 2 TNFα antagonists. Participants without prior failure or intolerance to biologics are not eligible. Participants who discontinued TNFα antagonist therapy for reasons other than failure or intolerance (eg, pregnancy) may be eligible after discussion with the medical monitor.

   Note: After the interim analysis, participants with inadequate response, loss of response, or intolerance to conventional UC therapy without prior exposure to biologics may be enrolled if deemed appropriate. Participants who discontinued biologics for reasons other than failure or intolerance (eg, pregnancy) may be eligible after discussion with the Medical Monitor.
7. If using corticosteroids must be on a stable dose of oral corticosteroids up to a maximum of 40 mg daily of prednisone or 9 mg daily of budesonide, or equivalent for at least 2 weeks prior to screening endoscopy and must be willing to follow a mandatory taper of corticosteroids from enrollment.

Exclusion Criteria:

Gastrointestinal Exclusion criteria:

1. Has any of the following UC-related complications:

   1. Acute severe UC.
   2. The participant has had extensive colonic resection, subtotal or total colectomy.
   3. The participant has clinical evidence of abdominal abscess or toxic megacolon.
   4. The participant has an ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine.
   5. Short bowel syndrome.
2. Has Crohn's colitis, indeterminate colitis, ischemic colitis, nonsteroidal anti-inflammatory drug (NSAID) induced colitis, idiopathic colitis (i.e, colitis not consistent with UC), radiation colitis, microscopic colitis, colonic mucosal dysplasia, or untreated bile acid malabsorption. Participants with a history of colonic mucosal dysplasia are also excluded.
3. Has uncontrolled primary sclerosing cholangitis.

Infectious Disease Exclusion Criteria:

1. Has any evidence of an active systemic infection during screening. Participants with nonsystemic infections (eg, active fungal infection of nail beds) may be eligible, if in the opinion of the investigator, inclusion of the participant will not interfere with the collection or interpretation of study results and poses no risk to the participant.
2. Has active or latent tuberculosis (TB), regardless of treatment history, as evidenced by any of the following:

   1. History of TB.
   2. A diagnostic TB test performed during screening that is positive, as defined by:

   i. A positive QuantiFERON test or 2 successive indeterminate QuantiFERON tests or ii. A tuberculin skin test reaction ≥10 mm (≥5 mm in subjects receiving the equivalent of >15 mg daily prednisone).
3. A positive test for hepatitis B virus (HBV).
4. A positive test for hepatitis C virus (HCV).
5. Evidence of, or treatment for, Clostridium difficile infection or other intestinal pathogen within 28 days prior to first dose of study treatment. Participants who test positive for C. difficile or other intestinal pathogens at screening and receive treatment may be enrolled or rescreened (if required) following confirmation of infection resolution.
6. Evidence of active Cytomegalovirus (CMV) infection at screening.

Medication exclusion criteria:

1. Has received immunomodulators (eg, 6-mercaptopurine, azathioprine, and methotrexate) within 4 weeks prior to first dose or immunosuppressants (eg, cyclosporine, tacrolimus) within 8 weeks prior to first dose.
2. Any medicinal product, herbal medication, or natural health product which might interfere with cytochrome P450 genotype 3A4 (CYP3A4) within 2 weeks prior to enrollment, except for any CYP3A4 modulator used to treat a C. difficile or an intestinal pathogen infection at screening.
3. Has received any of the following medical therapies for UC:

   1. IV antibiotics within 8 weeks prior to enrollment.
   2. Any rectal therapy for treatment of UC within 2 weeks prior to screening endoscopy.
   3. Chronic NSAID use defined as daily use for >2 consecutive weeks (Note: occasional use [<2 consecutive weeks] of NSAIDs and acetaminophen [<100 mg daily] for headache, arthritis, myalgias, or menstrual cramps and chronic low dose aspirin use [81-162.5 mg daily] for cardiovascular prophylaxis are permitted).
4. Has received a live virus or live bacterial vaccine within 4 weeks prior to enrollment or planned vaccination during the study and for 12 weeks after last dose.

General Exclusion Criteria:

1. Has any of the following cardiovascular or thrombotic conditions:

   1. Recent (within past 6 months) cerebrovascular accident, myocardial infarction, or coronary stenting.
   2. Recent (within past 6 months) moderate to severe congestive heart failure (New York Heart Association class III or IV).
   3. Prior history of thrombotic events, including deep vein thrombosis and pulmonary embolism.
   4. Known inherited conditions that predispose to hypercoagulability.
2. History of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy and/or splenomegaly.
3. A surgical procedure requiring general anesthesia within 3 months prior to screening or is planning to undergo major surgery during the study period.
4. Any investigational procedure ≤4 weeks prior to screening that, in the investigator's opinion, may interfere with interpretation of study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2027-07-09 (Estimated); Study Completion 2027-07-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Clinical Remission at Week 8 Based on Complete Mayo Score | At Week 8
  Clinical remission based on complete Mayo Score is where a participant achieves complete Mayo Score ≤2 points with no individual subscore >1 at Week 8. The complete Mayo Clinic Score includes 4 variables: Stool frequency, rectal bleeding, a Physician's Global Index (PGA) and Mayo endoscopic findings (MES). Each variable is scored on a 4-point scale (0-3 points) where 0=none and 3=severe disease and summed to give a total disease activity score (range, 0-12), with higher scores representing more severe disease activity.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Clinical Remission at Week 52 Based on Complete Mayo Score | At Week 52
  Clinical remission based on complete Mayo Score is where a participant achieves complete Mayo Score ≤2 points with no individual subscore >1 at Week 8. The complete Mayo Clinic Score includes 4 variables: Stool frequency, rectal bleeding, a Physician's Global Index (PGA) and Mayo endoscopic findings (MES). Each variable is scored on a 4-point scale (0-3 points) where 0=none and 3=severe disease and summed to give a total disease activity score (range, 0-12), with higher scores representing more severe disease activity.
Percentage of Participants Achieving Clinical Remission at Weeks 8, 14, and 26 Based on Partial Mayo Score | At Weeks 8, 14 and 26
  Clinical remission based on complete Mayo Score is where a participant achieves complete Mayo Score ≤2 points with no individual subscore >1. Partial Mayo Score consists of 3 variables of the Mayo Clinic Score: stool frequency, rectal bleeding and PGA. Each variable is scored on a 4-point scale (0-3 points) where 0=none and 3=severe disease. These scores are summed to give a total score range of 0 to 9 where higher scores indicate maximum disease activity.
Percentage of Participants Achieving Clinical Response at Weeks 2, 6, 8, 14, 26 and 52 Based on Complete or Partial Mayo Score | At Weeks 2, 6, 8, 14, 26, and 52
  Clinical response based on complete Mayo Score is where a participant achieves a reduction in complete Mayo score of ≥3 points and ≥30% from Baseline or a partial Mayo score of ≥2 points and ≥25% from baseline, if the complete Mayo score was not performed at the visit with an accompanying decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point. The complete Mayo Clinic Score includes 4 variables: Stool frequency, rectal bleeding, a PGA and MES. Each variable is scored on a 4-point scale (0-3 points) where 0=none and 3=severe disease and summed to give a total disease activity score (range, 0-12), with higher scores representing more severe disease activity.
Percentage of Participants Achieving Clinical Remission at Week 8 and Week 52 Based on Modified Mayo Score | At Weeks 8 and 52
  Clinical remission based on modified Mayo Score is where a participant achieves component modified Mayo score of ≤2 with modified MES ≤1, rectal bleeding = 0, and stool frequency ≤1. Modified Mayo Score consists of 3 variables: stool frequency, rectal bleeding and MES. Each variable is scored on a 4-point scale (0-3 points) where 0=none and 3=severe disease. These scores are summed to give a total score range of 0 to 9 where higher scores indicate maximum disease activity.
Percentage of Participants With Durable Clinical Remission at Week 8 and Week 52 | At Week 8 and Week 52
  Durable clinical remission is defined as the clinical remission at Week 8 and Week 52. Clinical remission is defined as complete Mayo Score of ≤2 points and no individual subscore >1 point at Weeks 8 and 52. The complete Mayo Clinic Score includes 4 variables: Stool frequency, rectal bleeding, a PGA and MES. Each variable is scored on a 4-point scale (0-3 points) where 0=none and 3=severe disease and summed to give a total disease activity score (range, 0-12), with higher scores representing more severe disease activity.
Percentage of Participants Using Oral Corticosteroids at Baseline Achieving Clinical Remission at Week 8 | At Week 8
  Clinical remission is defined as complete Mayo Score of ≤2 points and no individual subscore >1 point at Week 8. The complete Mayo Clinic Score includes 4 variables: Stool frequency, rectal bleeding, a PGA and MES. Each variable is scored on a 4-point scale (0-3 points) where 0=none and 3=severe disease and summed to give a total disease activity score (range, 0-12), with higher scores representing more severe disease activity.
Percentage of Participants With Corticosteroid-Free Clinical Remission at Week 8 | At Week 8
  Corticosteroid-free clinical remission is where a participant achieves corticosteroid-free clinical remission at Week 8. Clinical remission is defined as complete Mayo Score of ≤2 points and no individual subscore >1 point at Week 8. The complete Mayo Clinic Score includes 4 variables: Stool frequency, rectal bleeding, a PGA and MES. Each variable is scored on a 4-point scale (0-3 points) where 0=none and 3=severe disease and summed to give a total disease activity score (range, 0-12), with higher scores representing more severe disease activity.
Percentage of Participants Using Oral Corticosteroids at Baseline Achieving Clinical Remission at Week 52 | At Week 52
  Clinical remission is defined as complete Mayo Score of ≤2 points and no individual subscore >1 point at Week 52. The complete Mayo Clinic Score includes 4 variables: Stool frequency, rectal bleeding, a PGA and MES. Each variable is scored on a 4-point scale (0-3 points) where 0=none and 3=severe disease and summed to give a total disease activity score (range, 0-12), with higher scores representing more severe disease activity.
Percentage of Participants With Corticosteroid-Free Clinical Remission at Week 52 | At Week 52
  Corticosteroid-free clinical remission is where a participant achieves corticosteroid-free clinical remission at Week 52, and was off corticosteroids at least 3 months prior to Week 52. Clinical remission is defined as complete Mayo Score of ≤2 points and no individual subscore >1 point at Week 8. The complete Mayo Clinic Score includes 4 variables: Stool frequency, rectal bleeding, a PGA and MES. Each variable is scored on a 4-point scale (0-3 points) where 0=none and 3=severe disease and summed to give a total disease activity score (range, 0-12), with higher scores representing more severe disease activity.
Percentage of Participants Achieving Clinical Response at Week 8 | At Week 8
  Clinical response based on complete Mayo Score is where a participant achieves a reduction in complete Mayo score of ≥3 points and ≥30% from Baseline with an accompanying decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point. The complete Mayo Clinic Score includes 4 variables: Stool frequency, rectal bleeding, a PGA and MES. Each variable is scored on a 4-point scale (0-3 points) where 0=none and 3=severe disease and summed to give a total disease activity score (range, 0-12), with higher scores representing more severe disease activity.
Percentage of Participants With Mucosal Healing Based on MES at Week 52 | At Week 52
  Mucosal healing is defined as MES ≤1 point at Week 52. MES is a subscale of the Mayo score, an instrument designed to measure disease activity of UC. The subscale is graded from 0 to 3 based on the findings on endoscopy were 0= Normal appearance of mucosa, 1=mild disease (erythema, decreased vascular pattern), 2=moderate disease (marked erythema, lack of vascular pattern, friability, erosions), 3=severe disease (spontaneous bleeding, ulceration). Higher scores indicate more severe disease.
Percentage of Participants With Histological Remission Based on Geboes Score at Week 52 | At Week 52
  Histological remission is defined as Geboes score <2 at Week 52. The Geboes score is a histological grading system for assessing histological disease activity in UC. The Geboes score evaluates 7 histological features. It consists of 6 grades (0-6). Each of the grades is divided into subgrades, based on the severity of tissue abnormalities or the extent of inflammatory cell infiltration. The Geboes score ranges from 0.0 to 5.4, and higher grades are indicative of more severe disease activity.
Change in C-Reactive Protein Levels (CRP) From Baseline | Baseline to Weeks 2, 6, 8, 14, 26, 42 and 52
  CRP is a useful marker of inflammation in participants with inflammatory bowel disease (IBD). In participants with UC, elevated CRP has been associated with severe clinical activity.
Change in Fecal Calprotectin Concentrations From Baseline | Baseline to Weeks 2, 6, 8, 14, 26, 42 and 52
  Fecal calprotectin is a biomarker for intestinal inflammatory activity.
Change in Inflammatory Bowel Disease Questionnaire (IBDQ) Score From Baseline | At Weeks 8, 26 and 52
  The IBDQ is an instrument used to assess quality of life in adult participants with inflammatory bowel disease (IBD). It includes 32 questions on 4 domains of Health-Related Quality-of-Life (HRQOL): Bowel Systems (10 items), Emotional Function (12 items), Social Function (5 items), and Systemic Function (5 items). Participants are asked to recall symptoms and quality of life from the last 2 weeks and rate each item on a 7-point Likert scale (1=worst to 7=best). A total IBDQ score is calculated by summing the scores from each domain; the total IBDQ score ranges from 32 to 224, with lower scores reflecting worse HRQOL. A positive change from Baseline indicates improvement.
Change in Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Score From Baseline | At Weeks 8, 26 and 52
  The FACIT-F is a validated, 13-item questionnaire to assess fatigue in participants with a variety of chronic illnesses, including participants with IBD. Items are rated on a 5-point Likert scale and the total score ranges from 0 to 52 with lower scores representing greater fatigue.
Number of Participants With Adverse Events (AEs), Adverse Events of Special Interest (AESIs) and Serious Adverse Events (SAEs) | Up to 76 Weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not the occurrence is considered related to the study intervention.
Number of Participants With Clinically Significant Change in Vital Signs From Baseline | Up to 76 Weeks
  Vital signs will include body temperature, respiratory rate, blood pressure (resting more than 5 minutes), and pulse (resting more than 5 minutes).
Number of Participants With Clinically Significant Physical Examination Findings | At Baseline and From Week 14 to Week 72
  A baseline physical examination (defined as the assessment before first dose of study medication) will consist of the following body systems: general appearance; HEENT (head, eyes, ears, nose, and throat); cardiovascular system; respiratory system; gastrointestinal system; dermatologic system; extremities; musculoskeletal system; nervous system; lymph nodes; and other. All subsequent physical examinations will assess clinically significant changes from the assessment prior to first dose examination.
Number of Participants With Markedly Abnormal Laboratory Values | Up to Week 76
  Standard laboratory tests will include clinical chemistry, hematology, coagulation and urinalysis.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (50):
- United States (41):
  - Digestive Health Specialsits, Dothan, Alabama
  - GI Alliance Sun City, Sun City, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Hoag Hospital Newport Beach, Newport Beach, California
  - Endoscopic Research Inc, Orlando, Florida
  - Alliance Clinical Research of Tampa, LLC, Tampa, Florida
  - Gastroenterology Consultants, P.C., Roswell, Georgia
  - University of Chicago Medicine, Chicago, Illinois
  - GI Alliance - Illinois Gastroenterology Group - Glenview, Glenview, Illinois
  - GI Alliance - Illinois Gastroenterology Group LLC - Gurnee, Gurnee, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - GI Alliance, Metairie, Louisiana
  - Tulane University, New Orleans, Louisiana
  - Capital Digestive Care - MGG Group - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Huron Gastroenterology Associates, P.C., Ypsilanti, Michigan
  - MNGI Digestive Health, PA, Plymouth, Minnesota
  - Mid-America Gastro-Intestinal Consultants, Kansas City, Missouri
  - BVL Clinical Research, Liberty, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Weill Cornell Medical College- New York Presbyterian Hospital, New York, New York
  - Digestive Health Partners, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio Gastroenterology group, Inc., Columbus, Ohio
  - Gastro Intestinal Research Institute of Northern Ohio, LLC., Westlake, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny Health Network, Wexford, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Rapid City Medical Center, LLP, Rapid City, South Dakota
  - GI Alliance - Digestive Health Associates of Texas, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - GI Alliance - Mansfield, Mansfield, Texas
  - Gastroenterology Research of San Antonio, LLC, San Antonio, Texas
  - Texas Digestive Disease Consultants (TDDC), Southlake, Southlake, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - GI Alliance - Webster, Webster, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Washington Gastroenterology- GIA, Bellevue, Washington
  - Washington Gastroenterology- GIA, Tacoma, Washington
- Canada (9):
  - Barrie GI Associates Inc., Barrie, Ontario
  - London Health Sciences Centre, London, Ontario
  - West GTA Endoscopy Inc., Mississauga, Ontario
  - Viable Clinical Research - North Bay, North Bay, Ontario
  - Toronto Immune and Digestive Health Institute Inc. (TIDHI), North York, Ontario
  - ABP Research Services Corp., Oakville, Ontario
  - Taunton Surgical Centre, Oshawa, Ontario
  - Toronto Digestive Disease Associates (TDDA) Inc., Vaughan, Ontario
  - The Research Institute of the McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/bfc3d28999a04bba?idFilter=%5B%22Vedolizumab-4054%22%5D